CLINICAL TRIAL: NCT01742533
Title: A Phase Ι/Π Study of Human Cord Blood Mononuclear Cells and Human Umbilical Cord Mesenchymal Stem Cells Transplantation Combined With Hormone Replacement Therapy in Patients With Premature Ovarian Failure
Brief Title: Stem Cell Therapy Combined Hormone Replacement Therapy in Patients With Premature Ovarian Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Beike Bio-Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BKCR-POF-1(Ⅰ)
Record Dates: First submitted 2012-11-26; First posted 2012-12-05 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Premature Ovarian Failure，
Keywords: Hormone Replacement Therapy，; Premature Ovarian Failure，; Stem Cell Therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group1 : HRT plus hUCMSCs treatment: (Experimental): Participants will be given HRT plus human cord mesenchymal stem cells transplantation with a 12 menstrual Cycle follow-up.
  Interventions: Biological: human umbilical cord mesenchymal stem cells
- Group 2: HRT plus hCBMNCs and hUCMSCs therapy (Experimental): Participants will be given HRT plus combination of hCBMNCs together with hUCMSCs transplantation with a 12 menstrual Cycle follow-up.
  Interventions: Biological: hUCMSCs and hCBMNCs
- Group3 : HRT plus hCBMNCs treatment: (Experimental): Participants will be given HRT plus human cord blood mononuclear cells transplantation with a 12 menstrual Cycle follow-up.
  Interventions: Biological: human cord blood mononuclear cells
- Group 4:Hormone Replacement Therapy (Experimental): Participants will be given conventional therapy only with a 12 menstrual Cycle follow-up.
  Interventions: Drug: Hormone Replacement Therapy

INTERVENTIONS:
Biological: human umbilical cord mesenchymal stem cells
  Arms: Group1 : HRT plus hUCMSCs treatment:
Biological: hUCMSCs and hCBMNCs
  Arms: Group 2: HRT plus hCBMNCs and hUCMSCs therapy
Biological: human cord blood mononuclear cells
  Arms: Group3 : HRT plus hCBMNCs treatment:
Drug: Hormone Replacement Therapy
  Arms: Group 4:Hormone Replacement Therapy

SUMMARY:
Premature ovarian failure (POF) refers the occurrence of amenorrhoea, elevated serum gonadotrophins and hypoestrogenism levels in female before the age of 40. It has important physical and psychological consequences/impact in those patients.

Premature ovarian failure (POF) is currently managed by non-physiological sex steroid regimens which are inadequate at optimizing uterine characteristics.

Human umbilical cord mesenchymal stem cells (hUCMSCs) and human cord blood mononuclear cells (hCBMNCs) have been shown to have the ability to modulate the immune response and enhance angiogenesis, suggesting the novel and promising therapeutic strategy for POF.

In this study, the safety and efficacy of hUCMSCs and hCBMNCs transplantation combined with Hormone Replacement Therapy will be evaluated in patients with Premature Ovarian Failure. Participants will be followed for an expected average of 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Between age 18- 39 years, Female only.
* Diagnosed with Premature Ovarian Failure，and currently receiving Hormone Replacement Therapy;
* Willing to sign the Informed Consent Form.

Exclusion Criteria:

* Fragile X chromosome.
* polycystic ovary syndrome.
* HIV+.
* Autoimmune disease, e.g. lupus erythematosus, multiple sclerosis.
* Severe pulmonary and hematological disease, malignancy or hypo-immunity.
* Currently undertaking other treatment that may affect the safety/efficacy of stem cells.
* Pregnancy or lactation
* Enrollment in other trials in the last 3 months. • Other criteria the investigator consider improper for inclusion.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-06 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Serum Level of follicle-stimulating hormone | 48 weeks after treatment

SECONDARY OUTCOMES:
Uterine and Ovary characteristics of B ultrasound， including Uterine/Ovarian size and Blood Flow | 48 weeks after treatment
Modified Kupperman Score | 48 weeks after treatment
Incidence of Adverse Events and Serious Adverse Events | 48 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China